CLINICAL TRIAL: NCT03517904
Title: Comparison of Intravascular Ultrasound-Guided vs. Angiography-guided Angioplasty and Dual-antiplatelet v. Triple-antiplatelet Therapy for Outcomes of Drug-coated Balloon in the Treatment of Femoropopliteal Artery Disease (IVUS-DCB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2015-0093
Record Dates: First submitted 2016-06-20; First posted 2018-05-08 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Femoropopliteal Artery Disease
Keywords: Femoropopliteal artery disease, drug-coated balloon, angioplasty, antiplatelet therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVUS-guided group (Experimental): Intravascular ultrasound-guided intervention group
  Interventions: Procedure: IVUS-guided angioplasty
- Angiography-guided group (Active Comparator): Angiography-guided intervention group
  Interventions: Procedure: Angiography-guided angioplasty

INTERVENTIONS:
Procedure: IVUS-guided angioplasty — Angioplasty using drug-coated balloon (DCB) will be performed in standard manner. IVUS evaluation will be performed before predilation and after DEB treatment. In cases of stent implantation, additional IVUS evaluation will be performed after stenting. All lesions will be predilated using a plain balloon with a diameter 1 mm smaller than vessel size. Selection of DCB diameter will be chosen on the basis of IVUS measurement. Implantation of stents will be left to the operator's decision after reviewing IVUS findings after the DCB treatment. Generally, in presence of ≥ 50% residual stenosis or flow limiting dissections, implantation of stents is recommended.
  Arms: IVUS-guided group
Procedure: Angiography-guided angioplasty — Angioplasty using drug-coated balloon (DCB) will be performed in standard manner. All lesions will be predilated using a plain balloon with a diameter 1 mm smaller than vessel size. Selection of DCB diameter will be chosen on the basis of angiogram. Implantation of stents will be left to the operator's decision after reviewing the angiogram after the DCB treatment. Generally, in presence of ≥ 50% residual stenosis or flow limiting dissections, implantation of stents is recommended.
  Arms: Angiography-guided group

SUMMARY:
* Prospective, randomized, controlled, multi-center study
* A total of 240 subjects with femoropopliteal artery disease will be included according to inclusion and exclusion criteria.
* Patients will be randomized in a 1:1 manner into IVUS-guided or angiography-guided intervention group.
* Second 1:1 randomization into dual antiplatelet therapy (aspirin + clopidogrel) or triple antiplatelet therapy (aspirin + clopidogrel + cilostazol) is optional
* All patients will be treated with drug-coated balloons (In.PACT Admiral) for femoropopliteal lesions.
* Bare metal self-expandable stents will be used in addition according to findings of IVUS or angiography such as severity of arterial dissection or residual stenosis.
* Patients will be followed clinically for 1 year after the procedure.
* Ankle-brachial index and Image study follow-up (Duplex US or CT angiography) will be performed at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Symptomatic peripheral artery disease:

  * Moderate or severe claudication (Rutherford category 2 or 3)
  * Critical limb ischemia (Rutherford category 4 or 5)
* Femoropopliteal artery disease (stenosis > 50%)
* ABI <0.9
* Patients with signed informed consent

Exclusion Criteria:

* Acute critical limb ischemia
* Severe critical limb ischemia (Rutherford category 6)
* Known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, cilostazol, or contrast agents
* Patients requiring oral anticoagulation using warfarin or NOAC
* Age > 85 years
* Severe hepatic dysfunction (> 3 times normal reference values)
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* LVEF < 40% or clinically overt congestive heart failure
* Pregnant women or women with potential childbearing
* Life expectancy <1 year due to comorbidity
* Previous bypass surgery or stenting in the target femoropopliteal artery
* Untreated inflow disease of the ipsilateral pelvic or femoropopliteal arteries (more than 50% stenosis or occlusion)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Procedures lesion stenosis degree | at 12 months
  Absence of restenosis >50% by Duplex ultrasound, CT angiography, or catheter-based angiography

SECONDARY OUTCOMES:
Survival free from target vessel revascularization | 12 months
  Survival free from repeat intervention or surgical treatment due to loss of patency at the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SJ, Kim TH, Lee JH, Ahn CM, Lee SH, Lee YJ, Kim BK, Hong MK, Jang Y, Park HW, Jang JY, Park JH, Kim SH, Im E, Park SH, Choi D, Ko YG; IVUS-DCB Investigators. Intravascular Ultrasound-Guided vs Angiography-Guided Drug-Coated Balloon Angioplasty in Patients With Complex Femoropopliteal Artery Disease. JACC Cardiovasc Interv. 2025 Mar 10;18(5):558-569. doi: 10.1016/j.jcin.2024.10.052. Epub 2025 Jan 22. PMID 39846915